CLINICAL TRIAL: NCT03884556
Title: Phase 1/1b Study of the Safety of TTX-030 as a Single Agent and in Combination With Pembrolizumab or Chemotherapy in Patients With Lymphoma or Solid Tumor Malignancies
Brief Title: TTX-030 Single Agent and in Combination With Immunotherapy or Chemotherapy for Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trishula Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TTX-030-001
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor; Lymphoma
Keywords: Cancer; Metastatic Solid Tumors; Advanced Solid Tumors; Relapsed/Refractory Lymphoma; Prostrate Cancer; Pancreatic Cancer; Monotherapy; Combination Therapy; CD39; Adenosine Pathway; Immunotherapy; Immuno-oncology; PD-1; Checkpoint Inhibitor; Nab-paclitaxel; Gemcitabine; Pembrolizumab; Docetaxel; Bladder Cancer; Lung Cancer
MeSH Terms: conditions — Lymphoma; Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Lung Neoplasms | interventions — pembrolizumab; Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1, Single Agent (Experimental): TTX-030
  Interventions: Drug: TTX-030
- Arm 2, Anti-PD-1 Combination (Experimental): TTX-030 plus pembrolizumab
  Interventions: Drug: TTX-030; Drug: Pembrolizumab
- Arm 4, Chemotherapy Combination (Experimental): TTX-030 plus gemcitabine plus nab-paclitaxel
  Interventions: Drug: TTX-030; Drug: Gemcitabine; Drug: nab paclitaxel

INTERVENTIONS:
Drug: TTX-030 — Variable dose and schedule
Drug: Pembrolizumab — Dose and schedule per standard of care
  Arms: Arm 2, Anti-PD-1 Combination
Drug: Gemcitabine — Dose and schedule per standard of care
  Arms: Arm 4, Chemotherapy Combination
Drug: nab paclitaxel — Dose and schedule per standard of care
  Arms: Arm 4, Chemotherapy Combination

SUMMARY:
This is a phase 1/1b study of TTX-030, an antibody that inhibits CD39 enzymatic activity, leading to accumulation of pro-inflammatory adenosine triphosphate (ATP) and reduction of immunosuppressive adenosine, which may change the tumor microenvironment and promote anti-tumor immune response.

This trial will study the safety, tolerability, pharmacokinetics, and anti-tumor activity of TTX-030 as a single agent and in combination with an approved anti-PD-1 immunotherapy and standard chemotherapies.

ELIGIBILITY:
Abreviated Inclusion Criteria

1. Advanced solid tumor malignancy or relapsed/refractory lymphoma, or

   * eligible to receive single-agent pembrolizumab as standard of care, or
   * eligible to receive single-agent docetaxel as standard of care, or
   * advanced pancreatic adenocarcinoma and eligible to receive gemcitabine plus nab-paclitaxel as standard of care.
2. Age 18 years or older, is willing and able to provide informed consent
3. Evidence of measurable disease
4. Life expectancy > 12 weeks and Eastern Cooperative Oncology Group (ECOG) performance status of 0-1

Abbreviated Exclusion Criteria

1. History of allergy or hypersensitivity to study treatment components. Patients with a history of severe hypersensitivity reaction to any monoclonal antibody.
2. Use of investigational agent within 28 days prior to the first dose of study treatment and throughout the study
3. Receiving high-dose systemic steroid therapy or any other form of immunosuppressive therapy
4. History of severe autoimmune disease
5. Uncontrolled intercurrent illness or other active malignancy requiring ongoing treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - UC Irvine Cancer Center, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Nebraska Cancer Center Oncology Hematology West P.C., Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - West Cancer Center and Research Institute, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - Huntsman Cancer Intitute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: TTX-030 0.5 mg/kg: Participants in Arm 1 Escalation were administered IV 0.5 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 1.5 mg/kg: Participants in Arm 1 Escalation were administered IV 1.5 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 3.0 mg/kg: Participants in Arm 1 Escalation were administered IV 3.0 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 6.0 mg/kg: Participants in Arm 1 Escalation were administered IV 6.0 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 10 mg/kg: Participants in Arm 1 Escalation were administered IV 10 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 20 mg/kg: Participants in Arm 1 Escalation were administered IV 20 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 40 mg/kg: Participants in Arm 1 Escalation were administered IV 40 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1 Expansion: TTX-030 40 mg/kg Load, 30 mg/kg Q3W: Participants in Arm 1 Expansion received TTX-030 IV loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W.
- Arm 2 (Safety Lead-in and Expansion), Combination: Participants in Safety Lead-in portion and Expansion of Arm 2 received TTX-030 IV loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W and pembrolizumab IV at a dose of 200 mg on Day 1 of each 21-day treatment cycle.
- Arm 4 (Safety Lead-In and Expansion): Participants in Safety Lead-in and Arm 4 received TTX-030 IV loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W and received gemcitabine 1000 mg/m^2 + nab-Paclitaxel 125 mg/m^2 Days 1, 8, and 15 every 28 days.
Period: Overall Study
Arm/Group | Arm 1: TTX-030 0.5 mg/kg | Arm 1: TTX-030 1.5 mg/kg | Arm 1: TTX-030 3.0 mg/kg | Arm 1: TTX-030 6.0 mg/kg | Arm 1: TTX-030 10 mg/kg | Arm 1: TTX-030 20 mg/kg | Arm 1: TTX-030 40 mg/kg | Arm 1 Expansion: TTX-030 40 mg/kg Load, 30 mg/kg Q3W | Arm 2 (Safety Lead-in and Expansion), Combination | Arm 4 (Safety Lead-In and Expansion)
Started | 1 | 2 | 2 | 4 | 3 | 3 | 6 | 8 | 13 | 14
Completed | 1 | 2 | 2 | 4 | 3 | 3 | 6 | 8 | 13 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Histologically confirmed diagnosis of unresectable or metastatic solid tumor malignancy, or relapsed/refractory lymphoma, for which all standard therapies had been previously given.
Groups:
- Arm 1: TTX-030 3.0 mg/kg: Participants in Arm 1 Escalation were administered IV 3 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 6.0 mg/kg: Participants in Arm 1 Escalation were administered IV 6 mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 10 mg/kg: Participants in Arm 1 Escalation were administered IV 10mg/kg dose of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1 Expansion: TTX-030 40 mg/kg Load/30 mg/kg Q3W: Participants in Expansion received TTX-030 IV loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W.
- Total: Total of all reporting groups
Arm/Group | Arm 1: TTX-030 0.5 mg/kg | Arm 1: TTX-030 1.5 mg/kg | Arm 1: TTX-030 3.0 mg/kg | Arm 1: TTX-030 6.0 mg/kg | Arm 1: TTX-030 10 mg/kg | Arm 1: TTX-030 20 mg/kg | Arm 1: TTX-030 40 mg/kg | Arm 1 Expansion: TTX-030 40 mg/kg Load/30 mg/kg Q3W | Arm 2 (Safety Lead-in and Expansion), Combination | Arm 4 (Safety Lead-In and Expansion) | Total
Number analyzed (Participants) | 1 | 2 | 2 | 4 | 3 | 3 | 6 | 8 | 13 | 14 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2 | 2 | 2 | 4 | 4 | 9 | 6 | 31
  >=65 years | 0 | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 4 | 8 | 25
Age, Continuous [Median (Full Range); unit: years] | 26 [26 to 26] | 73 [72 to 74] | 59.5 [54 to 65] | 63 [55 to 67] | 64 [48 to 76] | 59 [56 to 76] | 61.5 [56 to 77] | 64.5 [51 to 81] | 57 [44 to 73] | 66.5 [46 to 83] | 63.5 [26 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 3 | 3 | 1 | 2 | 5 | 6 | 10 | 34
  Male | 0 | 1 | 0 | 1 | 0 | 2 | 4 | 3 | 7 | 4 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 6
  White | 1 | 1 | 2 | 3 | 2 | 2 | 6 | 6 | 12 | 10 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 2 | 4 | 3 | 3 | 6 | 8 | 13 | 14 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any clinically significant AE that occurred during Treatment Cycle 1 that the Investigator or Sponsor considered as possibly or likely related to TTX-030 as a single agent, or the combination of TTX-030 and other agent(s), and met the following criteria: NCI CTCAE Version 5.0 Grade 5 event, Grade 4 hematological or Grade≥3 non-hematological toxicities, or Grade≥3 irAEs. Laboratory abnormalities that were asymptomatic and deemed not clinically significant were not regarded as DLTs.
  During Dose Escalation, each dosing cohort was completed through the DLT observation window before escalation was allowed within its arm. In each Safety Lead-in cohort, all participants were closely monitored for the occurrence of DLTs.
Time Frame: 1 cycle (each cycle is 21-28 days)
Population: All participants in the Dose Escalation cohorts who received 1 infusion during the treatment cycle and completed safety evaluations through the end of the DLT period or experienced a DLT before the end of the DLT period (ie, participants started Cycle 2 or experienced a DLT).
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: TTX-030 1.5 mg/kg: Participants in Arm 1: TTX-030 was administered IV 1.5 mg/kg of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 3.0 mg/kg: Participants in Arm 1: TTX-030 was administered IV 3.0 mg/kg of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 6.0 mg/kg: Participants in Arm 1: TTX-030 was administered IV 6.0 mg/kg of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 10 mg/kg: Participants in Arm 1: TTX-030 was administered IV 10 mg/kg of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 20 mg/kg: Participants in Arm 1: TTX-030 was administered IV 20 mg/kg of TTX-030 Q3W on the first day of each 21-day treatment cycle.
- Arm 1: TTX-030 40 mg/kg: Participants in Arm 1: TTX-030 was administered IV 40 mg/kg of TTX-030 Q3W on the first day of each 21-day treatment cycle.
Arm/Group | Arm 1: TTX-030 1.5 mg/kg | Arm 1: TTX-030 3.0 mg/kg | Arm 1: TTX-030 6.0 mg/kg | Arm 1: TTX-030 10 mg/kg | Arm 1: TTX-030 20 mg/kg | Arm 1: TTX-030 40 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Objective Response Rate (ORR) (Except for Arm 1 and 2 Expansion Cohorts, Where ORR Was a Primary Endpoint)
Description: Anti-tumor activity in subjects treated with TTX-030 as single agent or in combination with specified regimens
Time Frame: Through study completion, an average of 1 year
Population: Participants in the Safety Analysis Set who had at least 1 post baseline evaluable tumor assessment unless death or clinical progressive disease (PD) occurred before the first post baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm 1: TTX-030 0.5 mg/kg: Participants in Arm 1: TTX-030 was administered IV 0.5 mg/kg of TTX-030 Q3W on the first day of each 21-day treatment cycle.
Arm/Group | Arm 1: TTX-030 0.5 mg/kg | Arm 1: TTX-030 1.5 mg/kg | Arm 1: TTX-030 3.0 mg/kg | Arm 1: TTX-030 6.0 mg/kg | Arm 1: TTX-030 10 mg/kg | Arm 1: TTX-030 20 mg/kg | Arm 1: TTX-030 40 mg/kg | Arm 4 (Safety Lead-In and Expansion)
Number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 3 | 6 | 13
percentage of participants | 1 [0.0 to 97.5] | 2 [0.0 to 84.2] | 1 [0.0 to 97.5] | 3 [0.0 to 70.8] | 2 [0.0 to 70.8] | 3 [0.0 to 70.8] | 6 [0.0 to 45.9] | 30.8 [9.1 to 61.4]

3. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: PK parameters of serum TTX-030 by Arm and Dose - Cycle 1
Time Frame: Cycles 1-3 (each cycle is 21-28 days)
Population: Dose-Normalized PK Parameters of Serum TTX-030
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Cmax (μg/mL)
Groups:
- Arm 1: TTX-030 0.5 mg/kg: Participants in Arm 1 was administered IV 0.5 mg/kg dose of TTX-030 Q3W on the first day of each 21-day
- Arm 1: TTX-030 1.5 mg/kg: Participants in Arm 1 was administered IV 1.5 mg/kg dose of TTX-030 Q3W on the first day of each 21-day.
- Arm 1: TTX-030 3.0 mg/kg: Participants in Arm 1 was administered IV 3.0 mg/kg dose of TTX-030 Q3W on the first day of each 21-day.
- Arm 1: TTX-030 6.0 mg/kg: Participants in Arm 1 was administered IV 6.0 mg/kg dose of TTX-030 Q3W on the first day of each 21-day.
- Arm 1: TTX-030 10 mg/kg: Participants in Arm 1 was administered IV 10 mg/kg dose of TTX-030 Q3W on the first day of each 21-day.
- Arm 1: TTX-030 20 mg/kg: Participants in Arm 1 was administered IV 20 mg/kg dose of TTX-030 Q3W on the first day of each 21-day.
- Arm 1: TTX-030 40 mg/kg: Participants in Arm 1 was administered IV 40 mg/kg dose of TTX-030 Q3W on the first day of each 21-day.
- Arm 1 Expansion: TTX-030 40 mg/kg Load/30 mg/kg Q3W: Participants in Arm 1 Expansion received TTX-030 IV loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W.
Arm/Group | Arm 1: TTX-030 0.5 mg/kg | Arm 1: TTX-030 1.5 mg/kg | Arm 1: TTX-030 3.0 mg/kg | Arm 1: TTX-030 6.0 mg/kg | Arm 1: TTX-030 10 mg/kg | Arm 1: TTX-030 20 mg/kg | Arm 1: TTX-030 40 mg/kg | Arm 1 Expansion: TTX-030 40 mg/kg Load/30 mg/kg Q3W | Arm 2 (Safety Lead-in and Expansion), Combination | Arm 4 (Safety Lead-In and Expansion)
Number analyzed (Participants) | 1 | 2 | 2 | 4 | 3 | 3 | 6 | 8 | 13 | 13
Cmax (μg/mL) | 4.91 (0) | 25.9 (8.2) | 35.2 (6.4) | 79.3 (49.3) | 188 (13.8) | 190 (75.8) | 629 (47.6) | 694 (56.8) | 647 (50.5) | 487 (27.3)

4. Primary Outcome: Objective Response Rate (ORR) - Arm 1 and Arm 2 Expansion Cohorts
Description: Anti-tumor activity in subjects treated with TTX-030 as single agent or in combination with specified regimens
Time Frame: Through study completion, an average of 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 Expansion: TTX-030 40 mg/kg Load/30 mg/kg Q3W | Arm 2 (Safety Lead-in and Expansion), Combination
Number analyzed (Participants) | 7 | 11
percentage of participants | 7 [0.0 to 41] | 9.1 [0.2 to 41.3]

ADVERSE EVENTS:
Time Frame: Up to 30 days from the last dose of TTX-030, a maximum duration of 2 years of treatment
Description: Safety population = all participants who received at least one dose or any partial dose of TTX-030.
Arm/Group | Arm 1: TTX-030 0.5 mg/kg | Arm 1: TTX-030 1.5 mg/kg | Arm 1: TTX-030 3.0 mg/kg | Arm 1: TTX-030 6.0 mg/kg | Arm 1: TTX-030 10 mg/kg | Arm 1: TTX-030 20 mg/kg | Arm 1: TTX-030 40 mg/kg | Arm 1 Expansion: TTX-030 40 mg/kg Load/30 mg/kg Q3W | Arm 2 (Safety Lead-in and Expansion), Combination | Arm 4 (Safety Lead-In and Expansion)
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/2 | 1/2 | 1/4 | 1/3 | 2/3 | 3/6 | 1/8 | 4/13 | 7/14
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 1/2 | 1/4 | 1/3 | 0/3 | 4/6 | 2/8 | 6/13 | 4/14
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2 | 2/2 | 4/4 | 3/3 | 3/3 | 3/6 | 6/8 | 13/13 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: TTX-030 0.5 mg/kg (N=1) | Arm 1: TTX-030 1.5 mg/kg (N=2) | Arm 1: TTX-030 3.0 mg/kg (N=2) | Arm 1: TTX-030 6.0 mg/kg (N=4) | Arm 1: TTX-030 10 mg/kg (N=3) | Arm 1: TTX-030 20 mg/kg (N=3) | Arm 1: TTX-030 40 mg/kg (N=6) | Arm 1 Expansion: TTX-030 40 mg/kg Load/30 mg/kg Q3W (N=8) | Arm 2 (Safety Lead-in and Expansion), Combination (N=13) | Arm 4 (Safety Lead-In and Expansion) (N=14)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: TTX-030 0.5 mg/kg (N=1) | Arm 1: TTX-030 1.5 mg/kg (N=2) | Arm 1: TTX-030 3.0 mg/kg (N=2) | Arm 1: TTX-030 6.0 mg/kg (N=4) | Arm 1: TTX-030 10 mg/kg (N=3) | Arm 1: TTX-030 20 mg/kg (N=3) | Arm 1: TTX-030 40 mg/kg (N=6) | Arm 1 Expansion: TTX-030 40 mg/kg Load/30 mg/kg Q3W (N=8) | Arm 2 (Safety Lead-in and Expansion), Combination (N=13) | Arm 4 (Safety Lead-In and Expansion) (N=14)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 6 (6) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 4 (4)
Back pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Edema peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Muscular weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT03884556/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT03884556/SAP_001.pdf